CLINICAL TRIAL: NCT03348670
Title: Explore the Relationship Between Single Nucleotide Polymorphisms and Abiraterone Response and Toxicity in Patients With Prostate Cancer.
Brief Title: Pharmacogenomics IND Commercial SNP Clinical Study - Abiraterone and Single Nucleotide Polymorphisms
Acronym: Drugs-SNPs
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair (Industry)
Responsible Party: Sponsor-Investigator, Han Xu, M.D., Ph.D., FAPCR, Sponsor-Investigator, IRB Chair, M.D., Ph.D., FAPCR, Sponsor-Investigator, Medical Director, IORG Director, Medical Monitor, Safety Officer, IRB Chair, Medicine Invention Design, Inc
Organization: Medicine Invention Design, Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: IND 178620 Commercial; FWA00015357 (Registry Identifier: HHS, Human Protections Administrator); IRB00009424 (Registry Identifier: HHS, IRB); IORG0007849 (Registry Identifier: HHS, IORG); NPI - 1831468511 (Registry Identifier: HHS, Health Care Provider Individual); NPI - 1023387701 (Registry Identifier: HHS, Health Care Provider Organization); IND 178620 (Registry Identifier: FDA IND Commercial)
Record Dates: First submitted 2017-11-15; First posted 2017-11-21 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; PC; SNP; Oncology; Genetics; Pharmacogenomics; CYP
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Prednisone; bicalutamide

STUDY DESIGN:
Intervention Model Description: * The usual approach group
  * The study approach group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: No-placebo and random and double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Abiraterone - Usual (Experimental): * ZYTIGA - Abiraterone
  * Combined Chemotherapy
  * ZYTIGA - abiraterone acetate tablet, film coated plus prednisone tablet plus BICALUTAMIDE tablet
  * Usual Approach Group
  Interventions: Drug: Abiraterone - Usual
- Abiraterone - Study (Experimental): * China Import - Abiraterone
  * Combined Chemotherapy
  * China Import - abiraterone acetate tablet plus prednisone tablet plus BICALUTAMIDE tablet
  * Usual Approach Group
  Interventions: Drug: Abiraterone - Study

INTERVENTIONS:
Drug: Abiraterone - Usual — * Oral
  * Abiraterone Combined Chemotherapy
  Other Names: ZYTIGA - abiraterone acetate tablet, film coated plus prednisone tablet plus BICALUTAMIDE tablet for Oral
  Arms: Abiraterone - Usual
Drug: Abiraterone - Study — * Oral
  * Abiraterone Combined Chemotherapy
  Other Names: China Import - abiraterone acetate tablet plus prednisone tablet plus BICALUTAMIDE tablet for Oral
  Arms: Abiraterone - Study

SUMMARY:
The usual approach group, 300 double blind random group separated PC patients currently used the Combined Chemotherapy on ZYTIGA - abiraterone acetate tablet, film coated plus prednisone tablet plus BICALUTAMIDE tablet, it will try to look for the relationship between the Abiraterone therapeutic efficacy and the CYP17 SNP Genotyping, and the relationship between the Abiraterone therapeutic safety and the SULT2A1 SNP Genotyping, based on Oxford precisely sequencing drug targets' genes.

The study approach group, 300 double blind random group separated PC patients currently used the Combined Chemotherapy on China Import - abiraterone acetate tablet plus prednisone tablet plus BICALUTAMIDE tablet, it will try to look for the relationship between the Abiraterone therapeutic efficacy and the CYP17 SNP Genotyping, and the relationship between the Abiraterone therapeutic safety and the SULT2A1 SNP Genotyping, based on Oxford precisely sequencing drug targets' genes.

DETAILED DESCRIPTION:
1. Detect drug target whole gene precision sequence of everyone patient for all 600 recruited double blind prostate cancer patients.
2. Mutually compare everyone patient drug target whole gene precision sequence for a total of 600 recruited double blind prostate cancer patients.
3. Calculate drug target gene SNPs in all 600 recruited double blind prostate cancer patients.
4. Correlate everyone patient drug target gene SNP to everyone patient drug efficacy.
5. Correlate everyone patient drug target gene SNP to everyone patient drug safety.
6. Mutually compare the usual approach group SNPs (300 double blind random group separated prostate cancer patients) with the study approach group SNPs (300 double blind random group separated prostate cancer patients).
7. Confirm the relationship between drug target gene SNPs and drug efficacy.
8. Confirm the relationship between drug target gene SNPs and drug safety.

ELIGIBILITY:
* Select 600 localized Prostate Cancer Patients without prostate resection
* Dosage Duration at least 90 days
* The usual approach group - Recruit 300 double blind random group separated prostate cancer patients currently used the Combined Chemotherapy on ZYTIGA - abiraterone acetate tablet, film coated plus prednisone tablet plus BICALUTAMIDE tablet, like as the usual approach group.
* The study approach group - Recruit 300 double blind random group separated prostate cancer patients currently used the Combined Chemotherapy on China Import - abiraterone acetate tablet plus prednisone tablet plus BICALUTAMIDE tablet, like as the study approach group.

Inclusion Criteria:

1. Clinical diagnosis of Prostate Cancer (PC)
2. Cancer in the prostate only
3. Prior therapy without orchiectomy
4. Prior therapy without prostate resection
5. Prior different chemotherapy must-need stop
6. Have no other cancer at the same time
7. Sign an informed consent form
8. Receive blood-drawing

Exclusion Criteria:

1. Treatment with other anti-cancer therapies and the therapies cannot be stopped currently
2. The patients with other serious intercurrent illness or infectious diseases
3. Have more than one different kind of cancer at the same time
4. Serious Allergy to Drugs
5. Serious Bleed Tendency
6. Serious Risks or Serious Adverse Events of the drug product label
7. Serious Risks or Serious Adverse Events of NCI Table of Side Effects
8. The prohibition of drug products
9. Have no therapeutic effects
10. Follow up to the most current label and plan for safety monitoring

Ages: 22 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate is male organ.
Enrollment: 600 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2026-05-18 (Estimated); Study Completion 2026-05-28 (Estimated)

PRIMARY OUTCOMES:
Measure and Report Abiraterone Drug Targets' SNP Genotypes which are effectiveness-associated, and which are risk-associated. | Up to 12 weeks
  * Recruit 300 double blind random group separated PC patients currently using the Combined Chemotherapy on ZYTIGA - Abiraterone tablet plus Prednisone tablet plus BICALUTAMIDE tablet to be the usual approach group.
  * Recruit 300 double blind random group separated PC patients currently using the Combined Chemotherapy on China Import - Abiraterone tablet plus Prednisone tablet plus BICALUTAMIDE tablet to be the study approach group.
  * Measure above every PC patient specific Abiraterone drug target (CYP17) SNP genotype in his or her WBC cell whole genome DNA with Oxford precisely sequencing.
  * Report every PC patient specific CYP17 SNP genotype in whole genome DNA sequence.
  * Measure above every PC patient specific Abiraterone drug target (SULT2A1) SNP genotype in his or her WBC cell whole genome DNA with Oxford precisely sequencing.
  * Report every PC patient specific SULT2A1 SNP genotype in whole genome DNA sequence.

CONTACTS AND LOCATIONS:
Overall Officials: HAN XU, MD/PhD/FAPCR, Study Chair — Medicine Invention Design, Inc. - IORG0007849 - NPI-1023387701; HAN XU, MD/PhD/FAPCR, Study Director — Medicine Invention Design, Inc. - IORG0007849 - NPI-1023387701; HAN XU, MD/PhD/FAPCR, Principal Investigator — Medicine Invention Design, Inc. - IORG0007849 - NPI-1023387701
Locations (1):
- Medicine Invention Design, Inc. - IORG0007849 - NPI-1023387701, Rockville, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FWA00015357 — http://ohrp.cit.nih.gov/search
- See also: IRB00009424 — http://ohrp.cit.nih.gov/search
- See also: IORG0007849 — http://ohrp.cit.nih.gov/search

DOCUMENTS (3):
  • Study Protocol (2023-08-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT03348670/Prot_006.pdf
  • Statistical Analysis Plan (2023-08-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT03348670/SAP_007.pdf
  • Informed Consent Form (2023-08-26): https://cdn.clinicaltrials.gov/large-docs/70/NCT03348670/ICF_008.pdf